CLINICAL TRIAL: NCT01955642
Title: Evaluation of the Biological Response to Clopidogrel in Patients With Ischemic Stroke : Role of Platelet alpha2-adrenergic Receptors
Brief Title: Evaluation of the Biological Response to Clopidogrel in Patients With Ischemic Stroke
Acronym: AAPIX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Groupe de Recherche sur la Thrombose (Other)
Responsible Party: Sponsor
Other Study IDs: 1208094; 2013-000313-20 (EudraCT Number)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Brain Ischemia; Ischemic Attack
Keywords: Clopidogrel; Brain Ischemia; Ischemic attack; Biological response to clopidogrel
MeSH Terms: conditions — Brain Ischemia | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AVC: Patients with non-cardioembolic AIC requiring initiation of treatment with clopidogrel as usual indications
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 75 mg milligrams per days of PLAVIX
  Other Names: PLAVIX(R)

SUMMARY:
Ischemic stroke (AIC) is the leading cause of non-traumatic disability in adults, the second leading cause of dementia and the third leading cause of death in France.

Clopidogrel is one of the recommended first line in the secondary prevention of AIC non cardioembolic origin. However recurrences occur in approximately 9% of patients receiving clopidogrel. Some studies in patients with coronary artery disease have made the connection between these treatment failures and non-biological response to clopidogrel. This non-biological response is found for approximately 30% to 50% of patients. Several mechanisms may explain this non-response. The most accepted mechanism is pharmacokinetic. Indeed, clopidogrel is a prodrug that requires intestinal absorption by P-glycoprotein (PGP) and a transformation by hepatic cytochrome into active metabolites. The genetic polymorphism of proteins involved in these two steps explain the low plasma concentration of active metabolites and thus the low efficacy of clopidogrel in some patients.

A new pharmacodynamic hypothesis suggests the involvement of platelet alpha 2-adrenergic receptors. The activation of these receptors potentiates signaling pathway P2Y12 receptor (channel inhibited by clopidogrel) and helps reduce platelet aggregation inhibiting response to clopidogrel.

DETAILED DESCRIPTION:
Interest in the biological response to clopidogrel in the AIC is innovative because few data are available in this area. In addition to testing a new pharmacodynamic hypothesis, we also wish to study and compare other measures of platelet function methods in order to be able to use commonly in treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Consent signed
* Patients with non-cardioembolic AIC requiring initiation of treatment with clopidogrel as usual indications
* normal standard biological tests

Exclusion Criteria:

* Need to continue aspirin therapy
* Patients with a recurrence of clopidogrel AIC
* Patient already tacking clopidogrel
* Drugs interfering with the adrenergic system alpha blockers, alpha 2 receptor agonists (alpha-methyldopa) and alpha2 receptor inhibitors (Mianserin, Mirtazapine, yohimbine)
* Contra indication of clopidogrel and / or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-cardioembolic AIC requiring initiation of treatment with clopidogrel as usual indications
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
adrenergic component of the platelet response | 5 days after taking clopidogrel
  adrenergic component of the platelet response is estimated by the difference between the maximum percentage of platelet aggregation by light transmission aggregometry (LTA) with the addition of ADP(adenosine diphosphate) + ADP versus selective agonist (epinephrine)

SECONDARY OUTCOMES:
VASP-CMF | After 5 days taking clopidogrel
  Platelet reactivity index (PRI) by VASP CMF (flow cytometry) method
ELISA VASP | After 5 days taking clopidogrel
  Platelet reactivity index (PRI-ELISA) using ELISA VASP
active metabolite of clopidogrel | After 5 days taking clopidogrel
  Rate of residual plasma active metabolite of clopidogrel (R-130964)
Genotyping of MDR-1 and P450 2C19 | After 5 days taking clopidogrel
  Genotyping of MDR-1 and P450 2C19

CONTACTS AND LOCATIONS:
Overall Officials: Jerome VARVAT, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France